CLINICAL TRIAL: NCT03164772
Title: A Phase 1/2 Study of Combination Immunotherapy and mRNA Vaccine in Subjects With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase 1/2 Study of Combination Immunotherapy and Messenger Ribonucleic Acid (mRNA) Vaccine in Subjects With NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Cancer Research Institute, New York City (Other); Boehringer Ingelheim (Industry); MedImmune LLC (Industry); CureVac (Industry); PharmaJet, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-012-VAC
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Non-small Cell Lung Cancer; NSCLC
Keywords: mRNA Vaccine; durvalumab; MEDI4736; anti-PD-L1; tremelimumab; anti-CTLA-4; BI 1361849; PharmaJet Tropis® device
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm A: BI 1361849 mRNA Vaccine + durvalumab (Experimental): The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Interventions: Drug: Durvalumab; Biological: BI 1361849; Device: PharmaJet Tropis® device
- Arm B: BI 1361849 mRNA Vaccine + durvalumab + tremelimumab (Experimental): The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; tremelimumab 75 mg was to be administered as an intravenous (IV) infusion every 4 weeks for the first 4 cycles (Arm B only); BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Biological: BI 1361849; Device: PharmaJet Tropis® device

INTERVENTIONS:
Drug: Durvalumab — anti-PD-L1
  Other Names: MEDI4736
Drug: Tremelimumab — anti-CTLA-4
  Arms: Arm B: BI 1361849 mRNA Vaccine + durvalumab + tremelimumab
Biological: BI 1361849 — mRNA Vaccine
  Other Names: CV9202
Device: PharmaJet Tropis® device — The PharmaJet Tropis® device was used for the intradermal administration of the BI 1361849 vaccine components.

SUMMARY:
This is an open-label, multicenter, 2-arm study to evaluate the safety and preliminary efficacy of the addition of a vaccine therapy to 1 or 2 checkpoint inhibitors for NSCLC.

Arm A: messenger ribonucleic acid (mRNA) Vaccine [BI 1361849 (formerly CV9202)] + anti-programmed death ligand 1 (PD-L1) antibody [durvalumab]

Arm B: messenger ribonucleic acid (mRNA) Vaccine [BI 1361849] + anti-programmed death ligand 1 (PD-L1) [durvalumab] + anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody [tremelimumab]

The run-in evaluation phase is followed by an expansion phase in which the cohort is expanded to 20 subjects (inclusive of subjects from the run-in).

DETAILED DESCRIPTION:
This was a Phase 1/2, open-label, multicenter, 2-arm study to evaluate the safety and preliminary efficacy of the addition of a vaccine therapy to 1 or 2 checkpoint inhibitors in subjects with NSCLC.

Up to 56 subjects were planned for enrollment from up to 8 clinical sites in 2 arms:

Arm A: mRNA Vaccine [BI 1361849 (formerly CV9202)] + anti-PD-L1 antibody [durvalumab]

Arm B: mRNA Vaccine [BI 1361849] + anti-PD-L1 [durvalumab] + anti-CTLA-4 antibody [tremelimumab]

Subjects must have had histologically confirmed metastatic NSCLC. For subjects with known EGFR or ALK/ROS-1 mutations, prior therapy must have included an EGFR tyrosine kinase inhibitor or ALK/ROS-1 inhibitor, respectively. Subjects may have had 1 prior line of anti-PD-1/PD-L1 therapy and must not have had progression at or before 12 weeks after start of the prior anti-PD-1/PD-L1 treatment.

ELIGIBILITY:
Inclusion Criteria

1. Histologic confirmation of metastatic NSCLC. For subjects with known EGFR or ALK/ROS-1 mutations, prior therapy must have included an EGFR tyrosine kinase inhibitor or ALK/ROS-1 inhibitor, respectively. Subjects may have had 1 prior line of anti-PD-1/PD-L1 therapy. Subjects who received prior anti-PD-1/PD-L1 therapy must have progressed during or after the prior anti-PD-1/PD-L1 therapy treatment, but not prior to Week 12 of treatment.
2. Measurable disease according to RECIST 1.1.
3. Availability of archival (diagnostic) specimens or willing to undergo a pre-treatment biopsy.
4. Subjects with treated brain metastases must have been treated with surgery and/or radiation therapy ≥ 21 days pre-study and must be clinically stable with no requirement for steroids.
5. Laboratory parameters for vital functions should be in the normal range.
6. ECOG Performance Status ≤ 2.
7. Body weight > 30 kg.

Exclusion Criteria

Subjects may not enter the study if they fulfill any of the following criteria:

1. Treatment with an investigational agent within 4 weeks of starting treatment or prior treatment with anti-CTLA-4 therapy.
2. Active, suspected or prior documented autoimmune disease, clinically significant cardiovascular disease, or clinically uncontrolled hypertension.
3. History of pneumonitis or interstitial lung disease, or any unresolved immune-related adverse events following prior therapy.
4. Major surgery within 4 weeks of starting treatment (or scheduled for surgery during the projected course of the study) or prior cancer vaccine treatment or allogeneic bone marrow transplantation.
5. Subjects who are immunosuppressed, including those with known immunodeficiency or have active infection or other serious illnesses.
6. Active infection including tuberculosis (TB), hepatitis B (HBV), hepatitis C, or human immunodeficiency virus (HIV). Subjects with a past or resolved HBV infection were eligible. Subjects positive for hepatitis C (HCV) antibody were eligible only if polymerase chain reaction was negative for HCV RNA.
7. History of severe allergic reactions to any unknown allergens or components of the study drugs.
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, bleeding disorders, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or serious chronic gastrointestinal conditions associated with diarrhea.
9. Subjects must not have donated blood while on study and for at least 90 days following the last durvalumab treatment or for 6 months after the last dose of tremelimumab (whichever was longer).
10. History of allogeneic organ transplant.
11. History of leptomeningeal carcinomatosis.
12. Active or prior malignancy except for history of other prior malignancy treated with curative intent which, in the opinion of the treating Investigator and the Sponsor, had minimal risk of interfering with safety or efficacy endpoints of the study.
13. Women of childbearing potential who were pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) or nursing.
14. Skin disease (e.g., psoriasis) that may prevent intradermal administration of the vaccine into the target areas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (5):
  - Research Facility, Gilbert, Arizona
  - Research Facility, Tampa, Florida
  - Research Facility, Detroit, Michigan
  - Research Facility, New York, New York
  - Research Facility, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST. Ann Oncol. 2014 Sep;25(suppl 4):iv361-iv72 [Abstract 4958]. doi: 10.1093/annonc/mdu342.23.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 subjects were enrolled; 24 into Arm A and 37 into Arm B. Of these 61 subjects, 57 were treated with at least one dose of study treatment; 23 in Arm A and 34 in Arm B.
  No dose adjustments were made and as a result all patients treated in each arm are presented.
Groups:
- Arm A: BI 1361849 mRNA Vaccine + Durvalumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  BI 1361849: mRNA Vaccine
- Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; tremelimumab 75 was to be administered as an intravenous (IV) infusion every 4 weeks for the first 4 cycles (Arm B only); BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  Tremelimumab: anti-CTLA-4
  BI 1361849: mRNA Vaccine
Period: Overall Study
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Started (Started is defined as started treatment.) | 23 | 34
Completed (Completed is defined as completed all 12 cycles of study treatment.) | 5 | 3
Not Completed | 18 | 31
Not completed — Death | 4 | 2
Not completed — Adverse Event | 1 | 4
Not completed — Progressive Disease | 11 | 21
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication.
Groups:
- Arm A: BI 1361849 mRNA Vaccine + Durvalumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  BI 1361849: mRNA Vaccine
- Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; tremelimumab 75 mg was to be administered every 4 weeks for the first 4 cycles (Arm B only); BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  Tremelimumab: anti-CTLA-4
  BI 1361849: mRNA Vaccine
- Total: Total of all reporting groups
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab | Total
Number analyzed (Participants) | 23 | 34 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.62) | 64.5 (11.76) | 64.7 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 24 | 34
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 31 | 47
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 14 | 28 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 23 | 34 | 57
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    PS 0 | 6 | 5 | 11
    PS 1 | 15 | 26 | 41
    PS 2 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.0 and classified by MedDRA system organ class (SOC) and preferred term. The severity was assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03. AEs were reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent was signed through 90 days after the last dose of study treatment. TEAEs are AEs that occurred or worsened in severity after administration of the first dose of study treatment.
  For each arm, the first 6 subjects were evaluated for dose limiting toxicities (DLTs).
  Deaths within the AE Reporting Period included all deaths that occurred during the study treatment period, or up to 90 days after the administration of the last dose of study drug or initiation of a new treatment.
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: BI 1361849 mRNA Vaccine + Durvalumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  BI 1361849: mRNA Vaccine
- Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose.The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; tremelimumab 75 mg was to be administered every 4 weeks for the first 4 cycles (Arm B only); BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  Tremelimumab: anti-CTLA-4
  BI 1361849: mRNA Vaccine
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
Participants
  Treatment-emergent Adverse Event (TEAE) | 23 | 33
  Treatment-related Adverse Event (TRAE) | 13 | 19
  Treatment-emergent Serious Adverse Event (SAE) | 14 | 22
  Treatment-related SAE | 1 | 3
  TEAE leading to treatment discontinuation | 5 | 8
  Deaths Within the AE Reporting Period | 5 | 7
  DLTs: number analyzed (Participants) | 6 | 6
  DLTs | 0 | 1

2. Secondary Outcome: Median PFS by RECIST 1.1 as Estimated Using the Kaplan-Meier Method
Description: Progression Free Survival (PFS) was measured from the date of the first dose of study treatment to the date of earliest disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or to the date of death, if disease progression did not occur. Per RECIST 1.1, progressive disease (PD) is defined as a ≥ 20% increase in the sum of the longest diameter of target lesions or the presence of new lesions.
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; tremelimumab 75 mg was to be administered as an intravenous (IV) infusion every 4 weeks for the first 4 cycles (Arm B only); BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  Tremelimumab: anti-CTLA-4
  BI 1361849: mRNA Vaccine
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
months | 2 [1.8 to 7.3] | 1.8 [1.2 to 2.8]

3. Secondary Outcome: Number of Subjects Without Progression at 8 and 24 Weeks by RECIST 1.1
Description: Progression-free Survival (PFS) was measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression did not occur. Per RECIST 1.1, progressive disease (PD) is defined as a ≥ 20% increase in the sum of the longest diameter of target lesions or the presence of new lesions.
Time Frame: up to 24 weeks
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: BI 1361849 mRNA Vaccine + Durvalumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose. The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  BI 1361849: mRNA Vaccine
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
Participants
  Number of Subjects Without Progression at Week 8 | 11 | 11
  Number of Subjects Without Progression at Week 24 | 8 | 3

4. Secondary Outcome: Median PFS by irRECIST as Estimated Using the Kaplan-Meier Method
Description: Progression-free Survival (PFS) was measured from the date of the first dose of study treatment to the date of earliest disease progression according to immune related Response Evaluation Criteria in Solid Tumors (irRECIST) or to the date of death, if disease progression did not occur. Per irRECIST, progressive disease (irPD) is defined as a ≥ 20% increase from nadir in the total measurable tumor burden (TMTB).
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
months | 2 [1.8 to 13.6] | 1.8 [1.2 to 2.8]

5. Secondary Outcome: Number of Subjects Without Progression at 8 and 24 Weeks by irRECIST
Description: Progression-free Survival (PFS) was measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression did not occur. Per irRECIST, progressive disease (irPD) is defined as a ≥ 20% increase from nadir in the total measurable tumor burden (TMTB).
Time Frame: up to 24 weeks
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
Participants
  Number of Subjects Without Progression at Week 8 | 11 | 11
  Number of Subjects Without Progression at Week 24 | 10 | 3

6. Secondary Outcome: Number of Subjects With Best Overall Tumor Response By RECIST 1.1
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up every 8 weeks starting 8 weeks after the last disease assessment. Per RECIST 1.1, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions or the presence of new lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study medication, had baseline and at least one post-baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 19 | 27
Participants
  CR | 0 | 0
  PR | 5 | 3
  SD | 7 | 8
  PD | 7 | 16

7. Secondary Outcome: Number of Subjects With Objective Responses at 8 and 24 Weeks By RECIST 1.1
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up every 8 weeks starting 8 weeks after the last disease assessment. Per RECIST 1.1, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions or presence of new lesions; stable disease (SD): small changes that do not meet above criteria. An Objective Response is defined as a CR or PR over a period of at least 4 weeks.
Time Frame: up to 24 weeks
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
Participants
  Week 8: Number of Subjects With an Objective Response | 5 | 0
  Week 8: Number of Subjects Without an Objective Response | 18 | 34
  Week 24: Number of Subjects With an Objective Response | 4 | 1
  Week 24: Number of Subjects Without an Objective Response | 19 | 33

8. Secondary Outcome: Duration of Response (DoR) By RECIST 1.1
Description: Duration of Response (DoR) was defined as the interval between the date of earliest determination of CR or PR to the date of earliest determination of progressive disease (PD), clinical progression or death, whatever occurred first.
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study medication, had baseline and at least one post-baseline tumor assessment and had a response of CR or PR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 5 | 3
weeks | 43.1 [24.1 to 53.5] | 25.1 [23.2 to 27.5]

9. Secondary Outcome: Number of Subjects With Best Overall Tumor Response By irRECIST
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up every 8 weeks starting 8 weeks after the last disease assessment. Per irRECIST, responses are categorized as follows: Complete Response (irCR): Complete disappearance of all target lesions; Partial Response (irPR): ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); Progressive Disease (irPD): ≥ 20% increase from nadir in TMTB; Stable Disease (irSD): not meeting above criteria.
Time Frame: up to 15 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 19 | 27
Participants
  irCR | 0 | 0
  irPR | 5 | 3
  irSD | 7 | 8
  irPD | 7 | 16

10. Secondary Outcome: Number of Subjects With Objective Responses at 8 and 24 Weeks By irRECIST
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up every 8 weeks starting 8 weeks after the last disease assessment. Per irRECIST, responses are categorized as follows: irCR: Complete disappearance of all target lesions; irPR: ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); irPD: ≥ 20% increase from nadir in TMTB; irSD: not meeting above criteria.
  An Objective Response is defined as an irCR or irPR over a period of at least 4 weeks.
Time Frame: up to 24 weeks
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
Participants
  Week 8: Number of Subjects With an Objective Response | 5 | 0
  Week 8: Number of Subjects Without an Objective Response | 18 | 34
  Week 24: Number of Subjects With an Objective Response | 4 | 1
  Week 24: Number of Subjects Without an Objective Response | 19 | 33

11. Secondary Outcome: Duration of Response (DoR) by irRECIST
Description: Duration of Response (DoR) was defined as the interval between the date of earliest determination of irCR or irPR to the date of earliest determination of progressive disease (irPD), clinical progression or death, whatever occurred first.
Time Frame: Up tp 15 months
Population: All subjects who received at least one dose of study medication, had baseline and at least one post-baseline tumor assessment and had a response of irCR or irPR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 5 | 3
weeks | 43.1 [24.1 to 53.5] | 25.1 [23.2 to 27.5]

12. Secondary Outcome: Median Overall Survival (OS) as Estimated Using the Kaplan-Meier Method
Description: After completion of treatment, all subjects were followed for survival every 6 months following initiation of study treatment until October 29, 2021 when all post-study follow-up was completed. OS was measured from the date of the first dose of study treatment to the date of death or last follow-up. Subjects lost to follow-up were censored on the date when they were last known to be alive.
Time Frame: up to October 29, 2021
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A: BI 1361849 mRNA Vaccine + Durvalumab: The BI 1361849 mRNA vaccine comprises 6 drug product components (F2408 coding for MUC1, F2409 coding for survivin, F2410 coding for NY-ESO-1, F2624 coding for 5T4, F2625 coding for MAGE-C2, and F2626 coding for MAGE-C1), which were provided and administered separately; each component was administered twice, thus there were 12 intradermal administrations of 100 µL (80 µg) each for each dose.The PharmaJet Tropis® device was used for the administration of the BI 1361849 components.
  Durvalumab 1500 mg was to be administered as an intravenous (IV) infusion every 4 weeks for 12 cycles; BI 1361849 was to be administered as 14 doses over the 12 cycles.
  Durvalumab: anti-PD-L1
  BI 1361849: mRNA Vaccine
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
Number analyzed (Participants) | 23 | 34
months | 23.5 [3.5 to NA] — Upper limit of confidence interval was not estimable due to small number of subjects with events. | 7.5 [3.4 to 10.5]

ADVERSE EVENTS:
Time Frame: up to 15 months All AEs occurring between the signing of informed consent and the off-study date (i.e., 90 days after the last dose of study treatment) are documented, regardless of the causal relationship to study drug. All cause mortality includes all deaths which were reported up until October 29, 2021.
Description: AEs that occur or worsen in severity after the first dose of study treatment are considered treatment emergent (i.e., TEAEs).AE documentation includes onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Arm A: BI 1361849 mRNA Vaccine + Durvalumab | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 12/23 | 22/34
Serious Adverse Events (participants affected / at risk) | 14/23 | 22/34
Other Adverse Events (participants affected / at risk) | 23/23 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: BI 1361849 mRNA Vaccine + Durvalumab (N=23) | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab (N=34)
Atrial flutter (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Lung infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Spine fracture (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stent placement (Surgical and medical procedures) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: BI 1361849 mRNA Vaccine + Durvalumab (N=23) | Arm B: BI 1361849 mRNA Vaccine + Durvalumab + Tremelimumab (N=34)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Palpitations (Cardiac disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 2
Vision blurred (Eye disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 11
Vomiting (Gastrointestinal disorders) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 8 | 11
Chills (General disorders) | 7 | 3
Pyrexia (General disorders) | 5 | 3
Oedema peripheral (General disorders) | 3 | 3
Injection site reaction (General disorders) | 1 | 4
Influenza like illness (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 2
Pain (General disorders) | 1 | 2
Axillary pain (General disorders) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 2
Lipase increased (Investigations) | 3 | 2
Weight decreased (Investigations) | 3 | 3
Amylase increased (Investigations) | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 2 | 2
Lymphocyte count decreased (Investigations) | 3 | 1
Weight increased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
The study was not randomized. There was disparity between the arms regarding the number of subjects treated before and after the protocol amendment which enabled inclusion of subjects who had 1 prior line of anti-PD-1/PD-L1 therapy. Seven subjects were treated in Arm A and 1 subject in Arm B before implementation of the amendment. The results for Arms A and B are not intended for comparison. All post study follow-up for the collection of survival was discontinued as of 29 October 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT03164772/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03164772/SAP_001.pdf